CLINICAL TRIAL: NCT02258750
Title: Experimental Study to Investigate the Effect of a High Fibre, Polydextrose-enriched Tomato Soup on Food Intake, the Experience of Appetite and Biomarkers of Satiation and Satiety
Brief Title: Assessing a Polydextrose Containing Soup on Food Intake, Appetite and Biomarkers of Satiation and Satiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of EU funding for the work package under investigation
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Dr. Una Masic, Post-Doctoral Associate, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ULKLSA002
Record Dates: First submitted 2014-09-25; First posted 2014-10-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Satiation, Satiety
MeSH Terms: interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polydextrose (Experimental): Tomato soup enriched with added polydextrose
  Interventions: Dietary Supplement: Polydextrose
- Control (Placebo Comparator): Tomato soup without added polydextrose
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Polydextrose — High fibre polydextrose enriched tomato soup (matched for sensory and nutritional characteristics to control) and eaten one hour before an ad-libitum lunch on study days. A 410g pre-packaged portion will be provided which contains 6% polydextrose compared to control.
  Arms: Polydextrose
Other: Control — Tomato soup (matched for sensory and nutritional characteristics to control) served in a 410g portion and eaten one hour before an ad-libitum lunch on study days.
  Arms: Control

SUMMARY:
This study will examine the impact of a soluble fibre (polydextrose) incorporated into a high fibre tomato soup on food intake (amount and choice), appetite ratings and biomarkers of satiation and satiety over 4-weeks. Specifically, the impact on the development of satiation within the fixed-load tomato soup containing the fibre, the development of satiety after the fixed-load meal containing fibre and intake at subsequent ad libitum meals will be examined as well as the insulin response and carbohydrate fermentation before and after 4-week dosing of the preload soup.

DETAILED DESCRIPTION:
The science underpinning both short (episodic) and long (tonic) term appetite regulation demonstrates that foods higher in macronutrients such as fibre can, under certain experimental conditions, produce great decreases in feelings of hunger and increases in fullness, post consumption, compared to equi-caloric loads of high carbohydrate or high fat. Given that fibre increases the release of GLP-1, slows down gastric emptying, prolongs nutrient absorption and, over long-term use increases the generation of short chain fatty acids (SCFAs) which have been linked to improved satiety responding, it is plausible that it will produce strong effects on within meal processes of satiation and satiety over the short- and long-term. Fibre has also been suggested to influence carbohydrate fermentation (via generation of these SCFAs) and improve the insulin response, additionally improving satiety. Ingredients may be added to boost fibre content such as the use of polydextrose, which is a non-digestible polysaccharide usually used as a dietary fibre in foods. Polydextrose has also been shown to increase levels of SCFAs due to its slow fermentation and has been related to reductions in subsequent intake and/or reduced hunger.

The aim of the current study is to assess the impact of a high fibre, polydextrose enriched tomato soup (experimental) or a low fibre tomato soup (control) on food intake, the experience of appetite and biomarkers of satiation and satiety.

Sample size: 86 males aged between 18 and 55 years with a body mass index (BMI) of between 23.0 and 28.0 kg/m2. A subset of 28 participants will undergo additional finger prick blood glucose and hydrogen breath test measures to assess biomarkers of satiation and satiety. Power calculations to ensure sufficient participants are included were based on power expected for a medium effect (0.25) at 80% power for a 2 condition between-measures design using G*power.

Methods: Participants will be invited to three full test day (baseline control, session 1; first dosing, session 2; one day prior to final dosing, session 3) sessions in which they will be provided with breakfast (tailored to individual resting metabolic rate (RMR) using the Schofield equation), the preload condition (receiving a high fibre polydextrose enriched or control tomato soup) one hour before an ad-libitum lunch and followed four hours later by an ad-libitum dinner and snack box. All test days will involve the use of standard operating proceedures. Pre-packaged portions of soup will be provided for a 4-week dosing period between study sessions 2 and 3 for all participants.

A subset of participants (N=28) will additionally undergo 3 further testing sessions (baseline control, session 0; second dosing, session 3; final dosing, session 4) in which a breakfast will be provided followed by the test product with additional glucose and carbohydrate fermentation measures collected for 3 hours before a light fixed portion meal.

Throughout test days participants will complete visual analogue scales (VAS) for appetite and palatability as well as questionnaires pertaining to eating behaviour and current sensations (including a gastrointestinal distress questionnaire).

Statistical analysis: Primary analysis will be comparison of subsequent ad-libitum energy intake between high fibre polydextrose enriched tomato soup compared to control using ANOVA and post-hoc tests. Meal duration and various appetite ratings will also be analysed as will biomarkers of satiety. The specified participant numbers (n=86) give an 80% probability of detecting an effect on energy intake.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 23-28 kg/m2
* Not dieting within the last month and not having lost significant amount of weight in the previous year.
* Not increased physical activity levels in the past 2-4 weeks or intending to modify them during the study
* Able to eat most everyday foods
* Breakfast eaters
* Soup consumers
* Written informed consent to be given

Exclusion Criteria:

* Those with significant health problems
* BMI < 23.0 kg/m2 or > 28.0 kg/m2
* Participants who self-report dieting currently or within the last month or having lost a significant amount of weight over the previous 6 months.
* Volunteers who have significantly changed their physical activity patterns in the past 2-4 weeks or who intend to change them during the study
* Gastrointestinal symptoms requiring treatment.
* Smokers or those who have recently ceased smoking (including electric cigarettes).
* Participants receiving systemic or local treatment likely to interfere with evaluation of the study parameters.
* Participants who work in the following areas: Nutrition, Dietetics, Food Research, Food Manufacturing or Supplements Industry.
* Participants currently adhering to any specific food avoidance diets such as Atkins, the South Beach diet or low Glycaemic Index (GI).
* Participants who have had bariatric surgery for weight control or other reason.
* Non breakfast eaters.
* Those reporting a history of anaphylaxis to food, significant general food allergies or specific allergies to any of the study foods.
* Participants with abnormal eating behaviour

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reductions in caloric intake at subsequent ad libitum meals after polydextrose-enriched soup intake | 90 minutes
  Calorie intake at ad-libitum lunch, dinner, and evening snack pack intake
More stable blood glucose response immediately after and after 4-week dosing of high fibre polydextrose enriched tomato soup compared to control | 180 minutes
  Finger prick blood glucose measures pre- (12:00pm), post-soup intake (12:15pm) and at 15 min and 30 min intervals for 3 hours post-intake (12:30pm, 12:45pm, 1:00pm, 1:30pm, 2:00pm, 2:30pm, 3:00pm, 3:30pm, 4:00pm, 4:30pm, 5:00pm)
Larger short chain fatty acid fermentation of carbohydrate after 4-week dosing of high fibre polydextrose enriched tomato soup compared to control | 180 minutes
  Hydrogen breath test measures pre- (12:00pm), post-soup intake (12:15pm) and at 15 min and 30 min intervals for 3 hours post-intake (12:30pm, 12:45pm, 1:00pm, 1:30pm, 2:00pm, 2:30pm, 3:00pm, 3:30pm, 4:00pm, 4:30pm, 5:00pm)

SECONDARY OUTCOMES:
Changes in subjective experience of satiation after ingestion of high fibre polydextrose enriched tomato soup compared to control | 30 minutes
  Visual Analogue Scale questionnaires (for appetite) completed before and after the soup and ad-libitum main meals. Questionnaire responses will be compared pre- and post-intervention across the 3 time points (Baseline day, Day 1 and final dosing day)
Changes in subjective experience of appetite and palatability in polydextrose tomato soup compared to control | 60 minutes
  Visual Analogue Scale questionnaires (for appetite and palatability taken before and after each meal (breakfast, soup, lunch, dinner) and at hourly intervals throughout the day. Questionnaire responses will be compared pre- and post-intervention across the 3 time points (Baseline day, Day 1 and final dosing day)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne A Harrold, Doctor, Principal Investigator — University of Liverpool; Jason CG Halford, Professor, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Background] Flood MT, Auerbach MH, Craig SA. A review of the clinical toleration studies of polydextrose in food. Food Chem Toxicol. 2004 Sep;42(9):1531-42. doi: 10.1016/j.fct.2004.04.015. PMID 15234083
- [Background] King NA, Craig SA, Pepper T, Blundell JE. Evaluation of the independent and combined effects of xylitol and polydextrose consumed as a snack on hunger and energy intake over 10 d. Br J Nutr. 2005 Jun;93(6):911-5. doi: 10.1079/bjn20051431. PMID 16022761
- [Background] Ranawana V, Muller A, Henry CJ. Polydextrose: its impact on short-term food intake and subjective feelings of satiety in males-a randomized controlled cross-over study. Eur J Nutr. 2013 Apr;52(3):885-93. doi: 10.1007/s00394-012-0395-4. Epub 2012 Jun 21. PMID 22717960
- [Background] Schwab U, Louheranta A, Torronen A, Uusitupa M. Impact of sugar beet pectin and polydextrose on fasting and postprandial glycemia and fasting concentrations of serum total and lipoprotein lipids in middle-aged subjects with abnormal glucose metabolism. Eur J Clin Nutr. 2006 Sep;60(9):1073-80. doi: 10.1038/sj.ejcn.1602421. Epub 2006 Mar 8. PMID 16523204